CLINICAL TRIAL: NCT05349240
Title: A Prospective, Single-arm, Multicenter Study to Evaluate the Efficacy and Safety of C2 CryoBalloonTM Ablation System in Patients With Esophageal Squamous Epithelium Dysplasia
Brief Title: C2 Esophageal Squamous Epithelium Dysplasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pentax Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBAS_DIII_19001
Record Dates: First submitted 2022-01-25; First posted 2022-04-27 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Esophageal Squamous Epithelium Dysplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Study Intervention (Experimental): All subjects will receive treatment with the study device.
  Interventions: Device: C2 CryoBalloonTM Ablation System.

INTERVENTIONS:
Device: C2 CryoBalloonTM Ablation System. — Cryoablation is used to ablate the tissue under the cryogenic condition. The device is mainly used to destroy the unhealthy tissues.

SUMMARY:
This study will evaluate the efficacy and safety of C2 CryoBalloonTM Ablation System for the cryoablation of dysplastic squamous tissue in patients with moderate to severe esophageal squamous epithelium dysplasia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of 18 to 80 years old (including 18 and 80 years old).
2. At least one unstained lesion (USL) in the esophagus upon high resolution upper gastrointestinal endoscopy with Lugol's staining. Flat (Paris type 0-IIb) USL, with the total area of one or more USLs having a maximum longitudinal size of 6 cm and covering a maximum of one-half of the esophageal circumference.
3. Patients with one or more biopsy confirmed esophageal squamous epithelium dysplasia areas within 6 months prior to enrollment, and the pathological diagnosis is moderate to severe esophageal squamous epithelium dysplasia.
4. No potential of lymph node metastasis by preoperative comprehensive evaluation.

Exclusion Criteria:

Inclusion criteria:

1. Male or female of 18 to 80 years old (including 18 and 80 years old).
2. At least one unstained lesion (USL) in the esophagus upon high resolution upper gastrointestinal endoscopy with Lugol's staining. Flat (Paris type 0-IIb) USL, with the total area of one or more USLs having a maximum longitudinal size of 6 cm and covering a maximum of one-half of the esophageal circumference.
3. Patients with one or more biopsy confirmed esophageal squamous epithelium dysplasia areas within 6 months prior to enrollment, and the pathological diagnosis is moderate to severe esophageal squamous epithelium dysplasia.
4. No potential of lymph node metastasis by preoperative comprehensive evaluation.
5. The patients are self volunteered to participate in the trial and will sign an informed consent form prior to enroll.

Exclusion criteria:

1. Females who are pregnant, lactating or plan to get pregnant during the study.
2. Known hypersensitivity to iodine.
3. Lesions within the target area such as: obvious ulcer; varices at risk of bleeding; active inflammation due to esophageal reflux into the treatment area; lesions view being not flat, or containing unfavourable unstained lesions (USLs) outside the designated treatment areas.
4. Esophageal stenosis preventing the passage of the endoscope to the treatment area. Esophageal stenosis or stricture preventing advancement of a therapeutic endoscope within 4 cm of the treatment area.
5. Having previously received Heller surgery: any previous ablative esophageal surgery (photodynamic therapy, multipolar electrical coagulation, argon plasma coagulation, laser treatment) or any previous esophageal surgery except for anti-reflux surgery.
6. Suffering from any cancer in the past 5 years.
7. Severe bleeding potential; patients on anti-coagulative therapy or stopping using anti-coagulative drugs for less than 7 days before enrollment or with impaired coagulation.

9) Patients with unstable vital signs 10) Anti-human immunodeficiency virus (HIV) antibody positive, both syphilis serology Treponema pallidum-specific antibody test and rapid plasma reagin positive.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who have complete remission of all the moderate to severe dysplasia in initial treatment area | 12 Month
  Percentage of complete remission at 12 months

SECONDARY OUTCOMES:
1) Percentage of subjects who have complete remission of all the moderate to severe dysplasia in initial by one time of treatment | 12 Month
  Percentage of patients who need only 1 treatment
2) Percentage of patients with complete remission of all the moderate to severe dysplasia in initial treatment area | 12 Month

OTHER OUTCOMES:
Safety Endpoints | 12 Months
  Frequency of adverse events and frequency of device related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Guiqi Wang, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (4):
- China (4):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Changzhi People's Hospital, Changzhi
  - The Second Hospital of Hebei Medical University, Shijiazhuang

IPD SHARING:
Plan to Share IPD: No